CLINICAL TRIAL: NCT04664816
Title: Chemopreventive Effect of Omega-3 Polyunsaturated Fatty Acids on the Recurrence of Non-Muscle Invasive Bladder Cancer: A Randomized, Double-Blinded, Placebo-Controlled Clinical Trial
Brief Title: Omega-3 Polyunsaturated Fatty Acids and Non-Muscle Invasive Bladder Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Elkashef, Assistant Lecturer of Urology, Urology and Nephrology Center, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Omega3-NMIBC
Record Dates: First submitted 2020-12-01; First posted 2020-12-11 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Non-Muscle Invasive Bladder Cancer
Keywords: Non-muscle invasive bladder cancer;; Transurethral resection of bladder tumor;; Omega-3 polyunsaturated fatty acids.
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- n-3PUFAs group (Experimental): These patients will receive omega-3 plus (1200 mg) orally, twice a day for at least 12 months. The treatment will start after TURBT, as soon as the histopathology will be obtained. The treatment will be discontinued if recurrence develops, unacceptable or serious adverse events occur or according to the patients' request.
  Interventions: Drug: n-3PUFAs Treatment
- Control group (Placebo Comparator): These patients will receive placebo orally, twice a day for at least 12 months. The treatment will start after TURBT, as soon as the histopathology will be obtained. The treatment will be discontinued if recurrence develops, unacceptable or serious adverse events occur or according to the patients' request.
  Interventions: Drug: Placebo Treatment

INTERVENTIONS:
Drug: n-3PUFAs Treatment — Omega-3 plus (1200 mg) orally, twice a day for at least 12 months.
  Other Names: Treatment
  Arms: n-3PUFAs group
Drug: Placebo Treatment — Placebo orally, twice a day for at least 12 months.
  Other Names: Control
  Arms: Control group

SUMMARY:
The investigators hypothesize that omega-3 polyunsaturated fatty acids (n-3 PUFAs) might have a role in prevention of the recurrence of non-muscle invasive bladder cancer (NMIBC).

The patients who are suffering from high-risk NMIBC will be randomly allocated into two groups: The first group (n-3 PUFAs group): 55 patients will receive omega-3 plus twice daily for one year after transurethral resection of bladder tumor (TURBT). The second group (Control group): 55 patients will receive placebo twice daily for one year after TURBT.

All patients will receive intravesical Bacillus Calmette-Guérin (BCG) immunotherapy and they will be followed up for two years.

The chemopreventive effect of n-3 PUFAs on the recurrence of NMIBC after TURBT will be studied via magnetic resonance imaging (MRI), inpatient cystoscopy, histopathological examination and molecular studies of the resected bladder tissues.

DETAILED DESCRIPTION:
The investigators hypothesize that omega-3 polyunsaturated fatty acids (n-3 PUFAs) might have a role in prevention of the recurrence of non-muscle invasive bladder cancer (NMIBC).

The patients who are suffering from high-risk NMIBC will be randomly allocated into two groups: The first group (n-3 PUFAs group): 55 patients will receive omega-3 plus (1200 mg) orally, twice a day for at least 12 months. The treatment will start after transurethral resection of bladder tumor (TURBT), as soon as the histopathology will be obtained. The treatment will be discontinued if recurrence develops, unacceptable or serious adverse events occur or according to the patients' request. The second group (Control group): 55 patients will receive placebo twice daily for one year after TURBT. Patients and care providers will be blinded to the medication given.

All patients will receive intravesical Bacillus Calmette-Guérin (BCG) immunotherapy and they will be followed up for two years.

The chemopreventive effect of n-3 PUFAs on the recurrence of NMIBC after TURBT will be studied via magnetic resonance imaging (MRI), inpatient cystoscopy, histopathological examination and molecular studies of the resected bladder tissues.

ELIGIBILITY:
Inclusion Criteria:

- Patients who are at high risk for recurrence of NMIBC after TURBT based on the following tumor characteristics:

* Stage Ta (G3, multifocal, or ≥ 2 occurrences within 12 months, including the current tumor),
* Stage T1 (any grade) and/or,
* Carcinoma in situ (CIS),
* Without any indication for radical cystectomy.

Exclusion Criteria:

- Patients with:

* ≥ T2 bladder cancer,
* Evidence of nodal metastasis,
* Associated upper tract urothelial carcinoma (UTUC) or
* Those who refuse.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Time to first recurrence. | 2 years
  Time to first recurrence is defined as the length of time from surgery to the first bladder recurrence or until last follow up.
Recurrence-free survival | 2 years
  Recurrence-free survival is defined as the length of time after treatment of non-muscle invasive bladder cancer that the patient survives without any radiological, histopathological, immunohistochemical or molecular evidence of tumor recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elkashef, Principal Investigator — Urology and Nephrology Center, Mansoura University, Egypt; Hassan Abol-Enein, Study Director — Urology and Nephrology Center, Mansoura University, Egypt; Ahmed A. Shokeir, Study Chair — Urology and Nephrology Center, Mansoura University, Egypt
Locations (1):
- Urology and Nephrology Center, Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No